CLINICAL TRIAL: NCT01688297
Title: Randomized Phase 1 Double-Blinded Placebo Controlled Trial to Determine the Safety and Immunogenicity of an Adenoviral-Vector Based Seasonal Influenza A Vaccine and dsRNA Adjuvant Administered Orally to Healthy Volunteers
Brief Title: Safety Study of an Oral Vaccine to Prevent Seasonal Influenza
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vaxart (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: VXA02-001 & VXA02-003
Record Dates: First submitted 2012-09-14; First posted 2012-09-19 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-05

CONDITIONS: Influenza
Keywords: Influenza; H1N1; flu; seasonal
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Low Dose VXA-A1.1 Oral Vaccine (Experimental): Two doses of replication incompetent adenovirus vaccine given in an oral tablet formulation.
  Interventions: Biological: VXA-A1.1 Oral Vaccine
- VXA Placebo Tablet (Placebo Comparator): Oral tablets of the same size and number as the vaccine tablet doses. Placebo arms were included during enrollment of each of the experimental dose groups to maintain the double-blind study design.
  Interventions: Biological: VXA Placebo Tablet
- Medium Dose VXA-A1.1 Oral Vaccine (Experimental): Two doses of replication incompetent adenovirus vaccine given in an oral tablet
  Interventions: Biological: VXA-A1.1 Oral Vaccine
- High Dose VXA-A1.1 Oral Vaccine (Experimental): One dose of replication incompetent adenovirus given in an oral tablet dose. This dose was studied under protocol VXA02-003.
  Interventions: Biological: VXA-A1.1 Oral Vaccine

INTERVENTIONS:
Biological: VXA-A1.1 Oral Vaccine — One or two doses of replication incompetent adenovirus oral tablet vaccine
  Other Names: Ad-HA-dsRNA (VXA-A1.1)
  Arms: High Dose VXA-A1.1 Oral Vaccine; Low Dose VXA-A1.1 Oral Vaccine; Medium Dose VXA-A1.1 Oral Vaccine
Biological: VXA Placebo Tablet — Off-white tablets similarly formulated to the active drug product tablets.
  Other Names: Placebo Control
  Arms: VXA Placebo Tablet

SUMMARY:
The purpose of this study was to demonstrate the safety and immunogenicity of an oral vaccine tablet to prevent seasonal influenza. The study was a placebo controlled, double blinded trial at a single site. The study was conducted under two separate protocols. Initially single administrations at two dose levels (low dose and mid dose) of the oral vaccine was tested in a placebo controlled study (37 subjects). And subsequently a single high dose of the oral vaccine was tested in a separate placebo-controlled study (24 subjects).

DETAILED DESCRIPTION:
Low and mid dose study was conducted under protocol number VXA02-001

High dose study was conducted under protocol number VXA02-003

ELIGIBILITY:
Inclusion Criteria:

* In good health as established by medical history, physical examination, and laboratory testing at the time of enrollment.

Exclusion Criteria:

* Positive for H1 influenza by HAI.
* Has had an influenza vaccine in the past 2 years.
* Current history of chronic alcohol consumption and/or illicit and/or recreational drug use.
* History of any confirmed or suspected immunodeficient or immunosuppressive condition
* Positive serology for HIV, HCV, or HBV
* Previous serious reactions to vaccination such as anaphylaxis, respiratory problems, hives, or abdominal pain.
* History of irritable bowel disease or other inflammatory digestive or gastrointestinal conditions that could affect the intended distribution of the vaccine targeting the mucosa of the small intestine
* Use of proton pump inhibitors(Nexium, Prilosec).
* Stool sample with occult blood at baseline exam

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2012-09; Primary Completion 2014-05 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Safety of an oral vaccine tablet as measured by reported solicited (reactogenicity) and unsolicited adverse events | One year following last vaccination

SECONDARY OUTCOMES:
Magnitude of humoral immune response to influenza as measured by functional assays | 28 Days and 180 Days post-vaccination
Magnitude of cellular immune responses to influenza as measured by functional assays | 28 Days and 180 Days post-vaccination

CONTACTS AND LOCATIONS:
Overall Officials: David Liebowitz, MD, PhD, Study Director — Vaxart, Inc.; Apinya Vutikullird, DO, Principal Investigator — WCCT
Locations (1):
- WCCT, Cypress, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Liebowitz D, Lindbloom JD, Brandl JR, Garg SJ, Tucker SN. High titre neutralising antibodies to influenza after oral tablet immunisation: a phase 1, randomised, placebo-controlled trial. Lancet Infect Dis. 2015 Sep;15(9):1041-1048. doi: 10.1016/S1473-3099(15)00266-2. PMID 26333337